CLINICAL TRIAL: NCT03430024
Title: Nuclear Myosin VI - a Therapeutic Target in Estrogen Receptor Positive Breast Cancer?
Brief Title: Nuclear Myosin VI - a Therapeutic Target in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maidstone & Tunbridge Wells NHS Trust (Other)
Collaborators: University of Kent (Other)
Responsible Party: Principal Investigator, Karina Cox, Consultant Breast and Oncoplastic Surgeon, Maidstone & Tunbridge Wells NHS Trust
Other Study IDs: 17/09/621_Myosin VI
Record Dates: First submitted 2018-01-11; First posted 2018-02-12 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Myosin VI; Estrogen receptor
MeSH Terms: conditions — Breast Neoplasms; Deafness, Autosomal Recessive 37 | interventions — Estrogen Receptor alpha

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: We will enrol 100 women who have been newly diagnosed with T2 (>2cm) palpable invasive breast cancer having primary surgical treatment at Maidstone Hospital. We will exclude all patients with a metabolic disorder, significant co-morbidities and locally advanced or metastatic disease as well as those with a previous history of cancer treatment. We will collect data on tumour size, grade and phenotype as well as ER, progesterone receptor (PR) and Her-2 expression status and patient demographic information.
  We will investigate the Association of Myosin VI with oestrogen receptor.
  Interventions: Other: Association of Myosin VI with oestrogen receptor
- Controls: A cohort of control breast tissue will be obtained from 20 patients undergoing benign surgical breast procedures. For those control patients having reduction mammoplasties the excised tissue will be core biopsied but patients having other types of benign surgery will have an extra core biopsy taken from breast tissue surrounding the lesion being excised.
  Interventions: Other: Association of Myosin VI with oestrogen receptor

INTERVENTIONS:
Other: Association of Myosin VI with oestrogen receptor — 1. Gene expression analysis - RNA will be extracted from 100mg of tissue and then subjected to RT-qPCR to determine the relative expression levels of several genes, including MVI and ER Targets. We will use the same approach to determine which isoforms of MVI are expressed in the tissue.
  2. Protein content analysis - Total protein will be extracted from 100 mg of tissue and western-blot analysis will be used to determine the relative amounts of MVI. Moreover, we will use cell fractionation to determine relative amounts of nuclear versus cytoplasmic protein.
  3. Genomic analysis - Chromatin-immunoprecipitation (ChIP) experiments we be performed upon 100 mg of tissue sample. Here we will determine the localisation of MVI on the genome within the different tissues.

SUMMARY:
Gene expression, the transfer of the genetic code into cellular proteins is one of the most fundamental processes in living cells. This process is orchestrated by protein-based molecular machines, called RNA polymerases that read the DNA sequence to generate messenger RNA (mRNA), which is translated by the cellular machinery to make proteins. Our cells have evolved elaborate regulation mechanisms to control these molecular machines and a breakdown in this regulation leads to diseases such as cancer.

Recently, molecules called myosins have been discovered in the genetic storage compartment of the cell (the nucleus) where they interact with RNA polymerases to regulate protein production. This is interesting because myosins are usually found outside the nucleus transporting cellular cargo or generating muscle contraction. In breast cancer cells, myosin is abundant and interacts with the oestrogen receptor. The majority of breast cancer in the UK is oestrogen receptor positive and activation of this receptor is an important factor controlling the growth of cancer cells. Oestrogen receptor activation appears to be dependent upon myosin and this research project will investigate how myosins are targeted to specific genes and how they are themselves regulated. This will greatly enhance our understanding of the role of nuclear myosins in oestrogen receptor positive breast cancer and may identify a novel therapeutic target for future drug development.

DETAILED DESCRIPTION:
Purpose and Design The primary aim of this project is to understand the significance of the newly discovered interaction between myosin VI (MVI) and the oestrogen receptor in breast cancer cells. The study will investigate the types of genes that MVI regulates and whether the sites of MVI - oestrogen receptor interactions (nucleus or cytoplasm) are important for the expression of oestrogen receptor targets. In breast cancer cells, oestrogen receptors can mutate to become permanently activated, leading to unrestrained tumour growth. Investigating the role of MVI in this metabolic scenario may reveal a potential therapeutic window for hormone refractory oestrogen receptor positive breast cancer.

In order to answer these questions, the methodology will use combination of experiments on established cell lines and patient samples.

The research proposal is a collaborative effort between Dr Chris Toseland (whose group has identified the link between MVI and the oestrogen receptor) at the University of Kent and the Breast Surgery, Pathology and Research and Development departments at Maidstone and Tunbridge Wells NHS Trust.

Recruitment Potential patients for recruitment will be identified at the weekly multi-disciplinary meeting following a diagnosis of primary breast cancer and a decision to proceed with surgery as the first treatment. The actual explanation of the study will take place during the first treatment planning consultation with the treating breast surgeon. The patient will be given written information about the study as well as a contact number of a research nurse/ breast care nurse specialist for them to call if they wish to be included in the study. A second clinic appointment will be made with the co-investigator Miss Karina Cox to re-discuss the trial and obtain written consent. The consultant surgeon is familiar with the process of consent and will determine whether the patient has capacity to give consent for the study. We will exclude all patients with a metabolic disorder, significant co-morbidities and locally advanced or metastatic disease as well as those with a previous history of cancer treatment as the results of the study may be affected by their underlying disorder, previous treatment or current medication.

Confidentiality The study will be conducted within the "Caldicott Principles'. Patients enrolled in the study will be given a unique identification number which will used on samples sent to The University of Kent for experiments. The clinical co-investigator will maintain a secure database of patient identifiable information including demographic and clinico-pathological tumour data.

Conflict of Interest There are no conflicts of interest with this study. Any publications relating to this research will be summarised and distributed to participating patients.

Tissue samples will not be stored indefinitely. All the tissue from the fresh frozen specimens will be used for the experiments. The paraffin slides, once analysed, will be returned from the University of Kent to Maidstone and Tunbridge Wells Pathology Department.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of early breast cancer
* Palpable tumour greater than 2cm
* Scheduled for primary surgical treatment

Exclusion Criteria:

* Locally advanced breast cancer
* Metastatic breast cancer
* Significant co-morbidities (ASA 4 or above)
* Past history of breast cancer

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tissue will be obtained from patients diagnosed with early invasive breast cancer undergoing primary surgery. We will enrol 100 women who have been newly diagnosed with T2 (>2cm) palpable invasive breast cancer having primary surgical treatment at Maidstone Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Gene expression of Myosin VI and oestrogen receptor targets in tumour tissue. | 24 hours
  RT-qPCR experiments to determine relative expression of Myosin VI and oestrogen receptor targets in tumour derived RNA and compare with control breast tissue.
Quantification of Myosin VI protein in tumour tissue. | 24 hours.
  Western-blot analysis and cell fractionation to determine relative amounts of Myosin VI compared to total protein extracted from 100mg of tumour tissue in nuclear and cytoplasmic compartments and compare with control tissue.
Localisation of Myosin VI on the tumour genome | 24 hours.
  Chromatin-immunoprecipitation experiments to determine the position of Myosin VI in the tumour genome and compare with control tissue.

SECONDARY OUTCOMES:
Comparison of nuclear Myosin VI and oestrogen receptor localisation between different breast cancer prognostic groups. | 3 months
  Immunohistochemisty experiments on paraffin preserved tumour tissue to determine the presence of nuclear Myosin VI and oestrogen receptors and, using a scoring system, compare between breast cancer prognostic groups and control tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Everest, Study Director — Maidstone and Tunbridge Wells NHS Trust
Locations (1):
- Maidstone and Tunbridge Wells NHS Trust, Maidstone, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vreugde S, Ferrai C, Miluzio A, Hauben E, Marchisio PC, Crippa MP, Bussi M, Biffo S. Nuclear myosin VI enhances RNA polymerase II-dependent transcription. Mol Cell. 2006 Sep 1;23(5):749-55. doi: 10.1016/j.molcel.2006.07.005. PMID 16949370
- [Background] Su AI, Welsh JB, Sapinoso LM, Kern SG, Dimitrov P, Lapp H, Schultz PG, Powell SM, Moskaluk CA, Frierson HF Jr, Hampton GM. Molecular classification of human carcinomas by use of gene expression signatures. Cancer Res. 2001 Oct 15;61(20):7388-93. PMID 11606367
- [Background] Dunn TA, Chen S, Faith DA, Hicks JL, Platz EA, Chen Y, Ewing CM, Sauvageot J, Isaacs WB, De Marzo AM, Luo J. A novel role of myosin VI in human prostate cancer. Am J Pathol. 2006 Nov;169(5):1843-54. doi: 10.2353/ajpath.2006.060316. PMID 17071605
- [Background] Wang H, Wang B, Zhu W, Yang Z. Lentivirus-Mediated Knockdown of Myosin VI Inhibits Cell Proliferation of Breast Cancer Cell. Cancer Biother Radiopharm. 2015 Oct;30(8):330-5. doi: 10.1089/cbr.2014.1759. Epub 2015 Sep 25. PMID 26407123 (Retraction: PMID 34596435 Cancer Biother Radiopharm. 2021 Dec;36(10):888)
- [Background] Yoshida H, Cheng W, Hung J, Montell D, Geisbrecht E, Rosen D, Liu J, Naora H. Lessons from border cell migration in the Drosophila ovary: A role for myosin VI in dissemination of human ovarian cancer. Proc Natl Acad Sci U S A. 2004 May 25;101(21):8144-9. doi: 10.1073/pnas.0400400101. Epub 2004 May 14. PMID 15146066
- [Background] Spudich G, Chibalina MV, Au JS, Arden SD, Buss F, Kendrick-Jones J. Myosin VI targeting to clathrin-coated structures and dimerization is mediated by binding to Disabled-2 and PtdIns(4,5)P2. Nat Cell Biol. 2007 Feb;9(2):176-83. doi: 10.1038/ncb1531. Epub 2006 Dec 24. PMID 17187061
- [Background] Morriswood B, Ryzhakov G, Puri C, Arden SD, Roberts R, Dendrou C, Kendrick-Jones J, Buss F. T6BP and NDP52 are myosin VI binding partners with potential roles in cytokine signalling and cell adhesion. J Cell Sci. 2007 Aug 1;120(Pt 15):2574-85. doi: 10.1242/jcs.007005. Epub 2007 Jul 17. PMID 17635994
- [Background] Naccache SN, Hasson T, Horowitz A. Binding of internalized receptors to the PDZ domain of GIPC/synectin recruits myosin VI to endocytic vesicles. Proc Natl Acad Sci U S A. 2006 Aug 22;103(34):12735-40. doi: 10.1073/pnas.0605317103. Epub 2006 Aug 14. PMID 16908842